CLINICAL TRIAL: NCT04918641
Title: Prospective, Natural History Study of Patients With Sanfilippo Syndrome Type A (MPS IIIA)
Brief Title: Natural History Observational Study of MPS IIIa in SMC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SMC-2020-10-164-003
Record Dates: First submitted 2021-04-28; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-04

CONDITIONS: Sanfilippo Syndrome A
MeSH Terms: conditions — Mucopolysaccharidosis III | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — CSF, urine, and serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No treatment: This is a longitudinal, prospective, observational, natural history study of patients with MPS IIIA to identify potential surrogate endpoints for future trials via standardized clinical, biochemical, neurocognitive, developmental, behavioral, and imaging measures.
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — Physical, developmental, neurological, behavioral, and neurocognitive assessments

SUMMARY:
To characterize the clinical course of mucopolysaccharidosis type IIIA (MPS IIIA), and identify potential endpoints for future treatment trials.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MPS IIIA
* Has the ability to comply with protocol requirements, in the opinion of the investigator

Exclusion Criteria:

* Patient's assent is unattainable, or the patient's parent(s), or patient's legally authorized representative(s) is/are unable to understand the nature, scope, and possible consequences of the study, or do/does not agree to comply with the protocol defined schedule of assessments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Initial patient eligibility is based on patient age and on a confirmed diagnosis of MPS IIIA.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-07-28 (Estimated); Study Completion 2024-07-28 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Bayley Scales of Infant Development-III/Kaufman Assessment Battery for Children-II (BSID-III/KABC-II) Age-Equivalent Scores | Baseline, 12 months, and 24 months
  The Bayley Scales of Infant and Toddler Development-Third Edition (BSID-III) is an individually administered test designed to assess the developmental functioning of infants and toddlers. The Bayley-III assesses development in five areas: cognitive, language, motor, social-emotional, and adaptive behavior. Children under the age of 3 will be tested for this. The Kaufman Assessment Battery for Children-Second Edition (KABC-II) is a clinical instrument for assessing cognitive development. Children over the age of 3 will be tested for this. Raw scores will be converted to age- equivalent scores to measure ability, skill, and knowledge, expressed as the age at which most individuals reach the same level (age norm; range: 0, unbound ). A positive value indicates improvement. The BSID-III and KABC-II age- equivalent scores will be based on the cognitive domain and average non-verbal age-equivalent score, respectively.
Change From Baseline in Vineland Adaptive Behavior Scales-II (VABS-II) Age-equivalent Scores | Baseline, 12 months, and 24 months
  The age equivalent score represents the age in months of the typical and normal individual who would achieve the same result as the one who was tested.
  The age equivalent scores are assessed by Vineland Adaptive Behavior Scales, Expanded Interview Form, Second edition (VABS-II). The Vineland is designed to measure the adaptive behavior of individuals from birth to age 90.
  The Vineland-II contains 5 domains each with 2-3 subdomains. The main domains are Communication, Daily Living Skills, Socialization, Motor Skills, and Maladaptive Behavior. A positive value indicates improvement in health and cognition.
Change from Baseline in MPS health Assessment Questionnaire, Sanfilippo Behavior Rating Scale | Baseline, 12 months, and 24 months
  Change from baseline in the SBRS scale assessed by parent report using the Sanfilippo Behavior Rating Scale form.

SECONDARY OUTCOMES:
Imaging characteristics | Baseline, 12 months
  MRI will be used to assess changes in the size of various organs affected by the disease, including the brain, liver, and spleen.
Echocardiography | Baseline, 6 months, 12 months, and 24 months
  2-D Echocardiography will be used to assess heart valve abnormalities and ventricular hypertrophy.
Hearing assessments | Baseline, 12 months, and 24 months
  The function of hearing will be assessed using Auditory Brainstem Response (ABR).
Sleep habits | Baseline, 12 months, and 24 months
  Patient sleep habits will be assessed using Children's Sleep Habits Questionnaire (CSHQ).
Ophthalmology assessments | Baseline, 12 months, and 24 months
  Change from Baseline in lens opacification
Change From Baseline in Quality of Life (ITQoL/PedsQL) Questionnaire | Baseline, 12 months, and 24 months
  Infant Toddler Quality of Life (ITQoL): The ITQoL Questionnaire is a generic, validated health status measure for children including items and scales to measure aspects of physical functioning, development, pain, mood, behavior, general health, and impact on parents. A positive value indicates improvement.
  Pediatric Quality of Life Inventory (PedsQL): Pediatric Quality of Life Inventory (PedsQL) is a modular approach to measuring health-related quality of life (HRQOL) in healthy children and adolescents and those with acute and chronic health conditions. Lower scores indicate better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: SungYoon Cho, Study Director — Samsung Medical Center